CLINICAL TRIAL: NCT04532450
Title: Outcomes of Fenestrated and Branched Stent Grafts to Treat Secondary Type 1 Endoleak After Endovascular Aneurysm Repair : A Prospective Multicentre Study
Brief Title: Outcomes of FEVAR and BEVAR to Treat Secondary Type 1 Endoleak After EVAR: A Prospective Multicentre Study
Status: Completed | Type: Observational
Sponsor: University Paul Sabatier of Toulouse (Other)
Responsible Party: Principal Investigator, Aurélien Hostalrich, Dr Aurelien Hostalrich, University Paul Sabatier of Toulouse
Other Study IDs: UPaulSabatierToulouse
Record Dates: First submitted 2020-07-09; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal aortic aneurysm; Failed EVAR; Type 1A endoleak; Fenestrated stent graft; EVAR
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Branched / fenestrated aortic stent graft — Endovascular repair of an aortic aneurysm with a branched/fenestrated stent graft to revascularise all visceral arteries together with exclusion of the aortic aneurysm.

SUMMARY:
Ten percent of the population above 60 years develops an aortic abdominal aneurysm. In case of rupture, this pathology leads to death in more than 70% of the cases.

Over the past ten years, Endovascular Aortic Aneurysm Repair (EVAR) has been the most used technique for elective treatment for abdominal aortic aneurysms (AAA) in patients with a favorable anatomy. But despite excellent postoperative results with a significant reduction of mortality , a close follow-up of these patients is mandatory to detect any potential endoleaks particularly in patients with a long-life expectancy.

Failed Endovascular Infrarenal Aortic Aneurysm Repair (EVAR) with development of a proximal endoleak exposes the patient to the risk of rupture and must be treated. This type of endoleaks are often related to dilatation of the proximal neck of the AAA, and of the suprarenal aorta, making the use of any aortic fixation system, or uncovered stent ineffective. In these cases, open surgical conversion with stent graft removal is possible but at the price of a significant morbidity and mortality.

The alternative is the use of a fenestrated or branched stent graft (F/BEVAR) extending the proximal sealing zone to a non-diseased aorta.

The goal of this study was to evaluate the technical feasibility, early and midterm outcomes of (F/BEVAR) in patients with a proximal endoleak following a standard EVAR.

The investigators performed a multicentre study between January 2010 and December 2019 in 8 French University Centres which included 85 patients with 3 years of post operative follow-up.

DETAILED DESCRIPTION:
Between January 2010 and December 2019, all patients (n=85) who developed after EVAR, a secondary type IA endoleak, and received a F/BEVAR stent graft were entered in a prospective multicentre study bringing together 8 French university centres.

Type IA secondary endoleak was defined as an endoleak appearing during follow-up, but absent on computed tomography angiography (CTA) within 30 days of EVAR. All aetiologies leading to the development of this endoleak were recorded in the study, including any abnormality of the infra-renal stent graft, any aneurysmal evolution of the neck of the infra-renal aneurysm, and any aneurysmal evolutionof the inter-renal or thoracoabdominal aorta.

All patients gave their informed consent for the operation. Following the European regulation on data management, the database was anonymised, upon completion.

All patients had a preoperative assessment of cardiac, renal, respiratory function and underwent an ASA physical status classification. All preoperative imaging were performed on <1.5 mm slices.

All F/BEVAR were performed using a COOK Zenith stent graft (Cook Medical Inc. Bloomington, Ind). The number of fenestrations used was based on the preoperative sizing made from 3D-CTA reconstructions. The investigators only used on-label F/BEVARs which were approved by the Zenith cook planning centre.

Procedures were performed under general, epidural or local anaesthesia, depending on the preference of the anesthesiologist, surgeon or patient. Procedures were performed in a conventional operating theatre or a hybrid room as described elsewhere.

General postoperative complications included any cause mortality. Acute kidney injury was defined following the KDIGO criteria , and myocardial infarction according to the generally accepted criteria. Postoperative respiratory complications were defined by the need for mechanical ventilation for more than 48 hours or re-intubation. SCI was classified according to the severity of the American Spinal Injury Association score and stroke was classified according to National Institute of Health Stroke Scale (NIHSS) .

The European Society for Vascular Surgery guidelines were used to define technical success, major adverse events, aneurysm sac changes, endoleak and device integrity .

F/BEVAR procedures were analysed in an intention to treat. A procedure was considered successful if the stent graft was implanted without any Type IA or type III endoleak, and with patent target arteries on peroperative angiography and on CTA or contrast enhanced ultrasound performed within the first week following the procedure. Target artery instability was defined as any branch-related death, rupture, occlusion or reintervention for stenosis, kink, endoleak, or disconnection. Monitoring during follow-up was carried out by CTA, at 3, 6 and 36 months thereafter. Any endovascular or open revision related to the procedure was recorded during follow-up.

Univariate analysis was performed using t-tests for normally distributed continuous variables, and Wilcoxon rank sum test for non-normally distributed continuous variables. Chi-square or Fisher tests was used when appropriate for categorical variables. Time dependent outcomes including patient survival, freedom from reintervention, freedom from endoleak and target arteries patency were reported using Kaplan-Meier time-to-event method. A p-value < .05 was used to assess statistical significance. All analyses were performed with SPSS V26, (IBM Corp.) and Medcalc ®.

ELIGIBILITY:
Inclusion Criteria:

* All patients who developed after primary endovascular aneurysm repair (EVAR), a secondary type IA endoleak, and received a Fenestrated stent graft as treatment
* All aetiologies leading to the development of this endoleak, any abnormality of the infra-renal stent graft, any aneurysmal evolution of the neck of the infra-renal aneurysm, and of the inter-renal or thoracoabdominal aorta.
* On-label Fenestrated gaft which were approved by the Zenith cook planning centre

Exclusion Criteria:

* Endovascular aortic repair<30 days
* Patients treated in emergency for aortic rupture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who developed more than 1 month after initial exclusion of an aortic abdominal aneurysm by a stent graft (EVAR) a proximal endoleak treated by a fenestrated stent graft to exclude a type 1A endoleak and to revascularise the renal arteries, the superior mesenteric artery and the celiac trunk.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of technical success | Up to 7 days following the procedure
  A procedure was considered successful if the fenestrated stent graft was implanted without any Type IA or type III endoleak, and with patent target arteries on peroperative angiography and on CTA or contrast enhanced ultrasound
Rate of general postoperative complications | Up to 31 days following the procedure
  Any cause mortality. Acute kidney injury defined by the KDIGO criteria, myocardial infarction, postoperative respiratory complications were defined by the need for mechanical ventilation for more than 48 hours or re-intubation. paraparesis or paraplegia according to the American Spinal Injury Association score and stroke according to National Institute of Health Stroke Scale (NIHSS) .
Rate of late complications | 36 months after the procedure
  Any complication occurring during follow-up.
Change in the aortic aneurysm diameter | 36 months after the procedure
  Aneurysm sac diameter: any change > 5 mm
Rate of unstable branches to target artery | 36 months after the procedure
  Any branch to target artery-related death, rupture, occlusion or reintervention for stenosis, kink, endoleak, or disconnection.
Rate of endoleak or F/B stent graft abnormality. | 36 months after the procedure
  Any endoleak, type IA, Type IB, Type II or any F/B stent graft abnormality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schermerhorn ML, Buck DB, O'Malley AJ, Curran T, McCallum JC, Darling J, Landon BE. Long-Term Outcomes of Abdominal Aortic Aneurysm in the Medicare Population. N Engl J Med. 2015 Jul 23;373(4):328-38. doi: 10.1056/NEJMoa1405778. PMID 26200979
- [Background] Katsargyris A, Yazar O, Oikonomou K, Bekkema F, Tielliu I, Verhoeven EL. Fenestrated stent-grafts for salvage of prior endovascular abdominal aortic aneurysm repair. Eur J Vasc Endovasc Surg. 2013 Jul;46(1):49-56. doi: 10.1016/j.ejvs.2013.03.028. Epub 2013 May 1. PMID 23642523
- [Background] Schanzer A, Beck AW, Eagleton M, Farber MA, Oderich G, Schneider D, Sweet MP, Crawford A, Timaran C; U.S. Multicenter Fenestrated/Branched Aortic Research Consortium. Results of fenestrated and branched endovascular aortic aneurysm repair after failed infrarenal endovascular aortic aneurysm repair. J Vasc Surg. 2020 Sep;72(3):849-858. doi: 10.1016/j.jvs.2019.11.026. Epub 2020 Mar 3. PMID 32144014
- [Background] Martin Z, Greenberg RK, Mastracci TM, Eagleton MJ, O'Callaghan A, Bena J. Late rescue of proximal endograft failure using fenestrated and branched devices. J Vasc Surg. 2014 Jun;59(6):1479-87. doi: 10.1016/j.jvs.2013.12.028. Epub 2014 Jan 29. PMID 24486036
- [Background] Goudeketting SR, Fung Kon Jin PHP, Unlu C, de Vries JPM. Systematic review and meta-analysis of elective and urgent late open conversion after failed endovascular aneurysm repair. J Vasc Surg. 2019 Aug;70(2):615-628.e7. doi: 10.1016/j.jvs.2018.11.022. Epub 2019 Apr 5. PMID 30956006
- [Result] Chaikof EL, Dalman RL, Eskandari MK, Jackson BM, Lee WA, Mansour MA, Mastracci TM, Mell M, Murad MH, Nguyen LL, Oderich GS, Patel MS, Schermerhorn ML, Starnes BW. The Society for Vascular Surgery practice guidelines on the care of patients with an abdominal aortic aneurysm. J Vasc Surg. 2018 Jan;67(1):2-77.e2. doi: 10.1016/j.jvs.2017.10.044. PMID 29268916
- [Derived] Hostalrich A, Mesnard T, Soler R, Girardet P, Kaladji A, Jean Baptiste E, Malikov S, Reix T, Ricco JB, Chaufour X; Association Universitaire de Recherche en Chirurgie (AURC). Prospective Multicentre Cohort Study of Fenestrated and Branched Endografts After Failed Endovascular Infrarenal Aortic Aneurysm Repair with Type Ia Endoleak. Eur J Vasc Endovasc Surg. 2021 Oct;62(4):540-548. doi: 10.1016/j.ejvs.2021.06.019. Epub 2021 Aug 5. PMID 34364770

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT04532450/Prot_SAP_000.pdf